CLINICAL TRIAL: NCT03013959
Title: Observation on Effect of Anti--inflammatory and Inhibition of Recurrence on the Herpes Simplex Keratitis After Topical NSAIDs Administration
Brief Title: Observation on the Herpes Simplex Keratitis
Acronym: OHSV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Yang Jiang, Attending Doctor，md, Peking Union Medical College
Other Study IDs: PekingUMC
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Keratitis, Herpetic
MeSH Terms: conditions — Keratitis, Herpetic | interventions — pyranoprofen

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Resting control group: The rest group is to study the effect of the inhibition of recurrence . Patients with redness, pain, decreased visual acuity and other reaction activity in the past 30 days are observed as control group
- Resting test group: The rest group is to study the effect of the inhibition of recurrence . Patients with redness, pain, decreased visual acuity and other reaction activity in the past 30 days are treated with pranoprofen and observed as test group
  Interventions: Drug: Pranoprofen
- Active control group: The active control group is to study the effect of anti--inflammatory. Patients with a new redness, pain, decreased visual acuity and other reaction activity recently are observed as control group
- Active test group: The active test group is to study the effect of anti--inflammatory. Patients with a new redness, pain, decreased visual acuity and other reaction activity recently are treated with pranoprofen and observed as test group
  Interventions: Drug: Pranoprofen

INTERVENTIONS:
Drug: Pranoprofen — it is an NSAIDs.As is reported, NSAIDs(pranoprofen) eye drops can suppress herpes simplex virus（HSV-1） reactivation and reduce inflammatory reaction in vitro and in vivo. In Clinical, there is no risk of corneal tissue melting, glaucoma, cataract by topical application of NSAIDs.
  Other Names: Pranopulin
  Groups: Active test group; Resting test group

SUMMARY:
As is reported, NSAIDs(pranoprofen ,bromfenac) eye drops can suppress herpes simplex virus（HSV-1） reactivation and reduce inflammatory reaction in vitro and in vivo. In Clinical, there is no risk of corneal tissue melting, glaucoma, cataract by topical application of NSAIDs. To explore more effective clinical treatment of viral keratitis patients to control the inflammatory damage, save the visual function and reduce the recurrence of the virus ,we observe the effect of anti-inflammatory and inhibition of recurrence on the herpes simplex virus after topical NSAIDs administration.

DETAILED DESCRIPTION:
Viral keratitis has now become the highest incidence and the most severe-caused blindness corneal disease in the worldwide, as is superior to bacterial keratitis and fungal keratitis. At present, clinical treatments mainly depend on local and systematic use of antiviral drugs for viral keratitis, which can inhibit replication of viruses in corneal tissues and directly damage viral action. However, basal studies for viral keratitis have suggested that pathological immune injury produced by the body also play an important role in the formation of corneal ulcer, the damage of visual function in patients, during the necrotic stromal inflammation phase, endotheliitis phase and even serious combination of iridocyclitis phase of viral keratitis. There is, however, a larger controversy in the hormone therapy for this disease clearly caused by pathological immune injury in medical world. Patients with infectious keratitis caused by viral infection, who receive hormone treatment, may cause viral replication enhanced and out of control, and hormone itself could also cause spontaneous corneal tissues fusion; hence, treatments combined with hormone have a certain risks. In clinical treatments, permanent corneal opacity caused by corneal inflammation responses will cause patients permanent visual acuity loss, after patients' corneal lesions were controlled with simple use of antiviral drugs. Another important reason is the high incidence of blindness caused by viral keratitis: herpesvirus, such as herpes simplex virus and herpes zoster virus, will involve trigeminal ganglia and hide after primary infection, and will repeatedly recur under the stimulation of excessive drinking, menstruation, taking a cold and operation etc.. Viral keratitis often does not cause patients severe visual impairment at initial onset. But, viruses in patients with herpes simplex virus keratitis show extremely high recurrence rates. As suggested in epidemiologic studies in the Euro-American countries, its recurrence rate could be up to 30% in the first year, and 46% in the second years. In most cases, transparent corneal tissues develop nephelium and even macular nebula opacities after repeated recurring, and patients eventually lose visual acuity, becoming people with blindness and disabilities. Nonsteroidal antiinflammatory drugs, such as pranoprofen and bromfenac sodium, show significant inhibition of virus recurrence and relief of corneal inflammation responses in experiments in vitro and animal experiments, which indicated in previous studies. In clinical, local application of nonsteroidal antiinflammatory drugs does not result in spontaneous corneal tissue fusion, drug-induced glaucoma, drug-induced cataract and other risks. In order to seek more effective clinical treatments for viral keratitis patients in terms of controlling inflammation injury, preserving visual functions and reducing virus recurrence, this study observed that pranoprofen, a nonsteroidal antiinflammatory drug, inhibits pathological immune injury of viral keratitis and prevents this disease recurring, according to the basal research background of viral keratitis.

ELIGIBILITY:
Inclusion Criteria:

1. Eyes with typical stromal infiltration, typical herpes simplex virus keratitis patients
2. Eyes with a history of recurrent erythema, pain, recurrent disease

Exclusion Criteria:

1. Patients with immune dysfunction or receiving immunosuppressive therapy
2. Patients with cardiac and pulmonary insufficiency
3. Patients with liver function, renal insufficiency
4. Patients with allergic reactions to related drugs
5. Patients with history of corneal surgery
6. Pregnant women and breast-feeding women
7. Patients with diabetes
8. Patients with malignant tumor history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Eyes with typical stromal infiltration, typical herpes simplex virus keratitis patients
  2. Eyes with a history of recurrent erythema, pain, recurrent disease
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
inhibition of recurrence on the herpes simplex virus | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, md, Study Director — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes